CLINICAL TRIAL: NCT05258019
Title: Prospective Clinical Study on Site Preservation of Alveolar Ridge After Tooth Extraction Before Dental Implantation
Brief Title: Site Preservation After Tooth Extraction
Status: Not yet recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2021-414
Record Dates: First submitted 2022-02-07; First posted 2022-02-28 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Osteogenesis Imperfecta; Total Absence of Permanent Teeth; Tooth Socket
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Geistlich Bio-Oss ® Particles + Bio-Gide ® collagen membrane: The first group of patients selected for site preservation will be performed with Bio-Oss ® Particles + Bio-Gide ® collagen membrane after tooth extraction
- Geistlich Bio-Oss ® Collagen + Bio-Gide ® collagen membrane: The second group of patients selected for site preservation will be performed with Bio-Oss ® Collagen + Bio-Gide ® collagen membrane after tooth extraction
- Conventional healing after tooth extraction, without site preservation: The third group of patients selected will be performed without site preservation after tooth extraction, and only conventional healing

SUMMARY:
This study is mainly targeted affected teeth which could not be retained, and patients are willing to undergo implant repair at the later stage. After teeth extraction, Geistlich Bio-Oss ® Particles or Bio-Oss ® Collagen are immediately implanted in the teeth extraction socket and covered with Bio-Gide ® collagen membrane for site preservation.Through postoperative follow-up, postoperative clinical and imaging objective indicators, combined with the subjective evaluation of surgeons and patients, and compared with conventional extraction treatment method, the study is aimed to evaluate the effectiveness of different site preservation of alveolar crest preservation, in order to reduce the alveolar bone width and height loss, effectively reduce alveolar bone absorption, or even achieve bone incrementation, thus to get the ideal site preservation effect, to improve the oral implant success rate, improve implant aesthetic score and patient satisfaction, provide more clinical standard reference of the clinical application of site preservation.

ELIGIBILITY:
Inclusion Criteria:

* patients willing to performed site preservation with Geistlich Bio-Oss ® Particles + Bio-Gide ® collagen membrane after tooth extraction;
* patients willing to performed site preservation with Geistlich Bio-Oss ® Collagen + Bio-Gide ® collagen membrane after tooth extraction;
* patients willing to performed no site preservation after tooth extraction and only conventional healing.

Exclusion Criteria:

* patients unwilling to sign the informed consent form and the letter of authorization;
* patients has a potential systematic diseases;
* patients had previously been treated with radiation therapy;
* patients can not re-visit on time.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who have teeth cannot be retained and are willing to do dental implant treatment at the teeth extration site.
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the alveolar crest height - central | up to 12 weeks after Dental extraction or site preservation surgery
  The central alveolar bone height of the ideal implant site will be measured with CBCT at 3 months after tooth extraction or plus site preservation
Changes in the alveolar crest width - central | up to 12 weeks after Dental extraction or site preservation surgery
  The central alveolar bone width of the ideal implant site will be measured with CBCT at 3 months after tooth extraction alone or plus site preservation

SECONDARY OUTCOMES:
Changes in the alveolar bone width - different depths | up to 12 weeks after Dental extraction or site preservation surgery
  The width of the alveolar bone at 1,3,5, and 7mm below the alveolar crest will be measured with CBCT at 3 months after tooth extraction or plus site preservation
Changes in the alveolar bone height - different horizontal sites | up to 12 weeks after Dental extraction or site preservation surgery
  The height of the alveolar bone will be measured at the mesial, central and distal of buccal and lingual of alveolar crest,and the midpoint of the mesial and distal of interproximal sites with CBCT at 3 months after tooth extraction alone or plus site preservation
Soft tissue thickness | up to 12 weeks after Dental extraction or site preservation surgery
  The thickness of soft tissue will be measured at middle, central, and distal sites of both buccal-lingual sides,3mm from free gingival margin
Plaque index (PLI) | up to 12 weeks after Dental extraction or site preservation surgery
  Each tooth extraction socket will be measured on 6 sites: buccal, central and lingual of both mesial-distal sides
Bleeding index (BI) | up to 12 weeks after Dental extraction or site preservation surgery
  Each tooth extraction socket will be measured on 6 sites: buccal, central and lingual of both mesial-distal sides
Probing depth (PD) | up to 12 weeks after Dental extraction or site preservation surgery
  Each tooth extraction socket will be measured on 6 sites: buccal, central and lingual of both mesial-distal sides
Phenotype assessment | up to 12 weeks after Dental extraction or site preservation surgery
  Whether thick or thin gingival biotype will be detected by the transparency of the soft tissue while periodontal probing diagnosis
Pain degree | up to 12 weeks after Dental extraction or site preservation surgery.
  The Visual Analogue Scale (VAS) pain score was evaluated: 0-10 (0: no pain; 1-3: slightly painful, acceptable; 4-6: painful, disrupt sleep, tolerable; 7-10: very painful, untolerable, affect sleep and diet)